CLINICAL TRIAL: NCT02614365
Title: Genes, Exercise, Neurocognitive and Neurodegeneration: Community-Based Approach
Acronym: GEMSII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Howard University (Other)
Collaborators: University of Southern California (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-MED-41E
Record Dates: First submitted 2015-03-24; First posted 2015-11-25 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise; Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental): 6-month 3-time/week aerobic exercise, and a 12-month passive follow-up.
  Interventions: Behavioral: Aerobic exercise
- Stretch Exercise (Active Comparator): 6-month 3-time/week stretch exercise, and a 12-month passive follow-up.
  Interventions: Behavioral: Stretch exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Cardiovascular fitness
  Arms: Aerobic Exercise
Behavioral: Stretch exercise — Muscle stretch
  Arms: Stretch Exercise

SUMMARY:
Whereas the advantageous effects of exercise-training on memory is increasingly recognized, the practicality and clinical usefulness of such interventions in community-dwelling older African Americans (AA)s Mild Cognitively Impaired (MCI) subjects, and the mechanism by which an effect occurs need elucidation. Because aerobic-exercise can improve emerging cardiovascular (CVD)-related risk factors for cognitive decline such as lipids, inflammatory cytokines and glucose homeostasis; the Investigators will examine training effects on these and related biomarkers. The imperative for this study is further underscored by the fact that, AAs: i) have high rates of dementia, and ii) have paucity of cross-sectional, and lack prospective data on the effects of exercise on cognition. To overcome barriers to recruitment and retention, enhance compliance with a long exercise program (3-times/week), and maximize the use of available resources, the Investigators will use a community-based approach. Therefore, the primary objectives of this study build on the Investigators' experience, and will compare the effects of aerobic-exercise to stretch-exercise (control) in community-dwelling AA MCI subjects. Following the initial 6 months active intervention, the aerobic-exercise group will follow a prescribed but free living 40 minutes, 3 time/week exercise regimen while the control group returns to usual care plus stretch-exercise for additional 12 months. This study will facilitate the estimation of sample size for a larger confirmatory study in AAs. A newly acquired direct oversight of the DC Ward-6 Senior Wellness Center and its infrastructures by the Howard University Division of Geriatrics will provide additional resources and access to the community. In addition to the Investigator's feasibility aims, the Investigators will determine performance on cognitive tasks using the Alzheimer's Disease Assessment Scale-Cognitive Sub-scale (ADAS-Cog) and Clinical Dementia Rating Scale (CDR) sum of boxes supplemented by tests of executive function (EF) and Functional Activity Questionnaire (FA) and together as ADAS-Cog-Plus; changes in brain volume regions of interest (ROI) with Magnetic Resonance Imaging (MRI), selected CVD and AD-related bio-markers.

DETAILED DESCRIPTION:
Although anticholinesterase therapies have greatly improved the symptomatic treatment of Alzheimer's disease (AD), they have not been demonstrated to significantly slow the disease progression; and amyloid-directed therapies have produced disappointing results. A promising evidence-based and relatively side-effect free lifestyle approach is emerging as an alternative or adjunct to drug therapy. In cross-section and prospective studies, and a few randomized controlled trials; aerobic exercise-training has been demonstrated to improve cognition in older subjects. However, the mechanisms of these effects remain poorly understood. Because it is now recognized that cardiovascular disease (CVD) risks can catalyze AD development, it is vital to test whether lifestyle adaptation shown to reduce CVD risks can favorably modify cognitive trajectories and markers of neurodegeneration. Such interventions may benefit those at an early and clinically discernible prodromal stage of AD such as mild cognitive impairment (MCI). Notably, such data are currently lacking in African Americans (AA)s who harbor higher rate of CVD risks and AD.

While a laboratory approach to exercise intervention study is required to prove causation, such a design may not lend itself to real-life application, and is demanding for many economically and educationally disadvantaged older AAs experiencing early symptoms of cognitive deterioration. To address this concern, the Investigators seek to initiate an 18-month study, testing real-life applicability of the effects of exercise adaptation on memory in a more ideal community setting. However, those who chose to exercise at an academic center will not be excluded. Collection of outcome measures at baseline, 3-month, 6-month, 9-month, 12-month and 18-month will provide pilot data to inform dose and duration effects of exercise on outcome measures. In addition to augmenting enrollments, the proposed approach will bolster retention.

The objectives of this pilot study, therefore, are to examine the feasibility of a community-based 18-month study (6-month active intervention and 12-month passive follow-up) aerobic exercise-training on neurodegeneration in AAs MCI subjects. The Investigators will test the hypotheses by randomizing subjects into one of 2 groups: 1.) aerobic-exercise; and 2.) stretch-exercise (control). The Investigators proposed that the aerobic-exercise group will perform better than control group on cognitive measures. Secondarily, the Investigators will determine whether training-induced changes in cognition relate to increases in brain volume. Exploratory, the Investigators will also investigate intervention effects on cerebrospinal fluid (CSF) biomarkers, selected CVD risk factors and biomarkers, cerebral oxygenation and Hypoxia-Inducible Factors (HIF-1α) gene expression, and Apolipoprotein E gene (APOE), to assess their mediation of training-induced changes in cognition.

A team of experienced Investigators in neuroimaging, neurology, cognitive neuroscience, and exercise physiology has been assembled to conduct this study. Working collaboratively with the District of Columbia Office on Aging (DCOA), the Directors of the Ward 6 Senior Wellness Center operated by DCOA, and the lead agencies on aging (community grassroots organizations supported by DCOA), the Investigators will recruit, enroll, randomize, and train participants at the wellness center. After obtaining informed consent and completing an initial assessment, participants will undergo initial exercise screening to determine their ability to exercise safely. Following randomization of 80 volunteers into aerobic-exercise (40) and control (40); baseline neuropsychological, neuroimaging and biomarker measurements will be obtained. Both groups will undergo 3 times/week supervised group-specific intervention at the wellness center for 6 months. After the initial 6 months of active intervention, the aerobic-exercise group will follow a prescribed but free living 40 minutes, 3 time/week exercise regimen, while the control group returns to usual care. Baseline tests will be repeated at 3 month, after 6 months (active intervention period); and at 9, 12 and 18 months (passive follow-up period). Treadmill, lumber puncture (LP) and brain magnetic resonance imaging (MRI) tests will occur only at baseline and 6 months. Between groups changes in cognitive performance, biomarkers, and neuroimaging measurements will be compared using appropriate multivariate methods.

While the Investigators remain cognizant of other planned or ongoing fitness and memory trial, the proposed study is unique in the sense that: it is a logical extension of the Investigators' ongoing work; tests the proposed hypotheses in predominantly AA sample in whom paucity of data remains, and therefore, will advance reduction in health disparity; will obtain data at multiple time-points (baseline, 3, 6, 9, 12 and 18 months) and therefore allow for the assessments of the effects of duration and dose of intervention on outcome measures; test the real-life applicability of the proposed intervention in a community setting; and generate pilot data on the mechanisms by which these interventions affects memory. Importantly, outcomes from this study may lead to practical and effective strategy to delay cognitive decline in populations at most risk, and can prevent or attenuate the physical, psychological and the economic burden associated with dementia in AAs.

ELIGIBILITY:
Main inclusion criteria:

* Age > 55 years
* Ability to exercise vigorously without causing harm to self
* Have Mild Cognitive Impairment (MCI) as defined under diagnosis above
* Have a study partner
* Be in good general health
* Willing to exercise for 12 months
* Willingness to undergo neuropsychological evaluation, PET scan of the brain, and have blood drawn

Exclusion Criteria:

* Age younger than 55 years
* Scored below 24 on the MMSE (have dementia)
* Have a Body Mass Index (BMI) ≥35,
* If a woman and peri-menopausal and unwilling to maintain current hormone replacement therapy status and allowed medication usage during the study.
* To avoid inaccurate HDL and HDL2-C determinations or avoid bias from familial hypercholesterolemia, respectively, participants with TG >400 mg/dl and those whose LDL-C levels >95% or HDL levels <10% of age and sex-adjusted norms will be excluded.
* Excluded medications: Medications with significant effect on memory such as anticholinergic (diphenhydramine, tricyclic antidepressants, benztropine); sedative hypnotics such as benzodiazepines; narcotics; and antiparkinsonian medications will all be excluded.
* Unstable medical conditions indicated by starting new medications within 6 weeks of enrollment will be disallowed.
* Concomitant Medication: Medications used in the therapy of AD (Reminyl, Aricept, Exelon, Namenda, Gingko Biloba) will be allowed if stable on these medications for 6 weeks prior to enrollment.
* Excluded Medical Diagnosis: To avoid misclassification bias, the Investigator will exclude persons with neurological, psychiatry or other clinical conditions likely to cause dementia. Participants having functional limitation preventing vigorous exercise, chronic disabling diseases, and alcoholism and drug abuse will be excluded.
* Clinically significant cerebrovascular disease including cortical infarct, strategically located subcortical gray matter or extensive white matter abnormalities.
* Treadmill screening exclusion criteria: include >2 mm ST depression, extra systole, chest pain, arrhythmias, hypotension and or dizziness or significant ST segment elevation during the treadmill test.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-07; Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessments | Change cognitive measures from baseline at 6 month
  Neuropsychological battery will be used to assess cognitive domains of interest.

SECONDARY OUTCOMES:
Brain MRI-derived regions of interest assessed by change in regions of interest brain volume | Change in regions of interest brain volume from baseline at 6 month and 12 month
  Brain MRI will be used as a screening tool and a measure brain volume
Cardiovascular disease-related markers and biomarkers assessed by change in lipids (mg/dl) | Change in lipids (mg/dl) from baseline at 3 month, 6 month, 9 month, 12 month and 18 month
  Cardiovascular disease related biomarkers.
Cardiovascular disease-related markers and biomarkers assessed by change in Nuclear Magnetic Resonance Spectroscopy measured lipids concentrations (nml/L) | Change in Nuclear Magnetic Resonance (NMR) Spectroscopy measured lipids concentrations (nml/L) from baseline at 3 month, 6 month, 9 month, 12 month and 18 month
  Cardiovascular disease related biomarkers.
Cardiovascular disease-related markers and biomarkers assessed by change in cytokines' levels (pg/ml) | Change in cytokines' levels (pg/ml) from baseline at 3 month, 6 month, 9 month, 12 month and 18 month
  Cardiovascular disease related biomarkers.
Alzheimer's disease-related markers and biomarkers assessed by change in serum levels of Tau (ng/L) and Abeta (ng/L) | Change in serum levels of Tau (ng/L) and Abeta (ng/L) from baseline to 3 month, 6 month, 9 month, 12 month and 18 month
  Cardiovascular disease and Alzheimer's disease related biomarkers.
Alzheimer's disease-related markers and biomarkers assessed by change in CSF levels of Tau (ng/L) and Abeta (ng/L) | Change in CSF levels of Tau (ng/L) and Abeta (ng/L) from baseline to 6 month.
  Cardiovascular disease and Alzheimer's Disease related biomarkers.
Cardiovascular disease and Alzheimer's disease-related gene-environment interactions. | Gene expression (fold change) from baseline at 3 month, 6 month, 9 month, 12 month and 18 month
  Cardiovascular disease and Alzheimer's disease related gene-environment interactions.
Alzheimer's disease-related markers and biomarkers and their gene-environment interactions. | Genotype at baseline
  Cardiovascular disease and Alzheimer's disease gene-environment interactions..
Number of participants enrolled | Number enrolled at baseline, and retained at 3 month, 6 month, 9 month,12 month and 18 month
  To test the feasibility of enrollment and retention of participants into a 6 month exercise study
Number of participants accepting of spinal tap procedure | Number of enrolled who had spinal tap at baseline and 6 month
  Acceptability of spinal tap procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Obisesan, MD, MPH, Principal Investigator — Howard University; Oyanumo Ntekim, MD, Study Director — Howard University
Locations (1):
- Howard University Clinical Research Unit, Washington D.C., District of Columbia, United States